CLINICAL TRIAL: NCT05870150
Title: The Development of a Non-typhoidal Salmonella Human Challenge Model: A Safety and Dose Escalation Study
Brief Title: Challenge Non-Typhoidal Salmonella (CHANTS) Study
Acronym: CHANTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: University of Oxford (Other); University of Liverpool (Other); PATH (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 21HH6989; 301659 (Other: IRAS Project ID); 21/PR/0051 (Other: REC reference)
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Salmonella Infections; Salmonella Typhimurium; Non-typhoidal Salmonella (NTS); Invasive Non-Typhoidal Salmonella Disease; Communicable Disease; Infections, Bacterial; Enteric Fever (Not Typhoid); Gastroenteritis
Keywords: Controlled human infection study; Human infection challenge model; Experimental human challenge
MeSH Terms: conditions — Salmonella Infections; Communicable Diseases; Bacterial Infections; Typhoid Fever; Gastroenteritis

STUDY DESIGN:
Intervention Model Description: A two-arm study where participants will receive one of two strains of Salmonella Typhimurium (ST19 or ST313).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ST19 (Experimental): Healthy volunteers will be challenged with Salmonella Typhimurium ST19
  Interventions: Biological: Salmonella Typhimurium
- ST313 (Experimental): Healthy volunteers will be challenged with Salmonella Typhimurium ST313
  Interventions: Biological: Salmonella Typhimurium

INTERVENTIONS:
Biological: Salmonella Typhimurium — Salmonella Typhimurium oral challenge. Dose-escalating (1-5x10^3 CFU, 1-5x10^4 CFU, 1-5x10^5 CFU, 1-5x10^6 CFU)

SUMMARY:
This protocol describes the challenge non-typhoidal Salmonella (CHANTS) study. This is a first-in-human phase 1, double-blinded, randomised, dose-escalation human infection study, conducted in healthy volunteers aged 18 to 50 years. The primary objective of the study is to perform a dose escalation with two strains (ST19 or ST313) to determine the infectious dose required for 60-75% of volunteers to develop Salmonellosis using a composite diagnostic criterion. The secondary objectives of the study are to describe and compare the clinical and laboratory features following controlled human infection. It is hoped that the successful establishment of an NTS human challenge model can be used in the future to test candidate vaccines for NTS disease.

DETAILED DESCRIPTION:
The overall aim of this study is to establish a controlled human infection model of invasive non-typhoidal Salmonella (iNTS) infection. The investigators will challenge healthy volunteers with two strains of Salmonella Typhimurium. Participants will be admitted to an inpatient quarantine facility after the challenge and treated with antibiotics when they meet defined criteria. The primary objective of the study is to perform a dose escalation to determine the infectious dose required for 60-75% of volunteers to develop Salmonellosis using a composite diagnostic criterion. The secondary objectives of the study are to describe and compare the clinical and laboratory features following controlled human infection with Salmonella Typhimurium. It is hoped that the successful establishment of an NTS human challenge model can be used in the future to test candidate vaccines for NTS disease.

Study design: Double-blinded randomised human infection study

Number of visits: 21 to 26 (depending on the outcome of the challenge)

Sample size: Up to 80 (depending on the outcome of the dose escalation study)

Study participants: Healthy adults aged 18 to 50 years inclusive

Challenge strain(s) Salmonella enterica subspecies enterica serovar Typhimurium strain 4/74 - Dose range from 1-5 x 10e1 to 1-5 x10e6 CFU suspended in sodium bicarbonate prior to oral ingestion. Produced to GMP.

Salmonella enterica subspecies enterica serovar Typhimurium strain D23580 - Dose range from 10e1-10e6 CFU suspended in sodium bicarbonate prior to oral ingestion. Produced to GMP.

Research procedures:

Screening Participants will complete an online questionnaire to assess their eligibility and provide information about their medical history. They may then be contacted by telephone to discuss any information they have provided or invited directly for a face-to-face appointment. The purpose of screening is to assess eligibility and provide an opportunity for the participant to be fully informed about the study and to ask any questions they may have.

At the screening visit, the study team will go through the study in detail and consent the participant to enrollment in the study.

If following the consent process the participant was willing to do so the study investigators would ask participants to complete a short quiz to ensure that the study had been understood and sign an informed consent form.

The study investigators will then ask questions about the participant's health, travel, medication and vaccination history, occupational and household contacts, undertake a physical examination including an ECG ('heart tracing') and take a urine and blood sample to assess eligibility.

Blood is screened for general health (to check a full blood cell count, kidney and liver function), HIV, hepatitis B and C, and coeliac disease as well as for a congenital immune deficiency that some people have without knowing (called IgA deficiency). Blood is also tested for the presence of the HLA-B27 gene which encodes for a protein called human leukocyte antigen B27 on the surface of white blood cells.

All participants are asked to complete a questionnaire to assess anxiety and depression. A separate questionnaire will be used to screen for symptoms of irritable bowel syndrome. In addition, participants are asked to attend a separate appointment for an abdominal ultrasound to check for gallstones and for aortic aneurysms,

For all females, the study investigators will perform a pregnancy test on their urine samples.

The study investigators will ask permission to contact the participant's GP to confirm eligibility and provide medical and vaccination records.

Once the results from these tests are received the study team will make an assessment of eligibility and this will be communicated to the participant. Once eligibility is confirmed then arrangements will be made for the challenge.

Enrollment The pre-challenge visit marks the start of formal enrolment in the study. This will take place one week before the challenge visit. At this visit, participants are asked to sign a second consent form to confirm that they are still willing to take part. The study investigators will check that there have been no changes to their health since the screening visit. The study investigators will also perform a brief medical examination and collect some extra tests, including blood, and urine. Will will give participants a kit to collect faecal samples to bring in at their next visit.

Challenge The day of the challenge is designated as Day 0. It marks the start of the busy study period. The challenge starts by admitting participants to our dedicated inpatient facility. Participants have a blood test taken and women would take a urine pregnancy test. Will also perform a lateral flow test for COVID-19. Participants are administered a sodium bicarbonate solution to neutralise stomach acid. This will be followed by a solution containing one of the two Salmonella Typhimurium strains. Participants will fast for a further 90 minutes after challenge.

After the challenge, participants are to remain as inpatients in quarantine for at least 7 days. Participants will be discharged when defined discharge criteria are met.

Discharge criteria

Participants will be discharged from the inpatient quarantine unit if the following criteria are met:

* Medically fit for discharge in the opinion of the study physician AND
* Complete resolution of diarrhoea (Bristol stool type 6-7) for 48 hours1 AND
* Seven days (168 hours) have elapsed since challenge

For patients diagnosed with Salmonellosis from day 0 to day 7, the following criteria apply:

* Antibiotic treatment has been initiated and patient has completed SD+96hrs follow up OR
* Resolution of Salmonella Typhimurium bacteraemia (if applicable)

After 7 days, participants will be allowed to leave the quarantine facility. They will continue to be seen in an outpatient setting for a further 7 days. At follow-up visits, diary entries will be reviewed, observations will be taken plus blood and stool samples.

Diagnosis and treatment After the challenge participants may develop symptoms of Salmonella infection or remain well. Participants may develop symptoms of Salmonella at any point after the challenge. The study investigaors might expect symptoms to start as soon as 12-48 hours after the challenge, but this can range from as short as 4 hours to as long as 3 days. Symptoms are expected to last between 3 to 7 days on average. If a participant develops pre-specified treatment criteria or invasive Salmonella infection the study investigators will start antibiotic treatment,

Treatment criteria

Antibiotics are commenced if ANY of the following apply:

* Any participant with Salmonella Typhimurium bacteraemia
* Fever ≥38oC for ≥12hrs
* Any participant with severe gastroenteritis
* Moderate gastroenteritis plus:

  * fever ≥38°C on one occasion and/or
  * ≥1 Grade 2 systemic symptoms
* Any participant with 3 or more of the following symptoms on the same day at Grade 2 or higher;

  * Headache
  * Fatigue/Malaise
  * Anorexia
  * Abdominal pain
  * Nausea
  * Vomiting
  * Myalgia
  * Arthralgia
  * Cough
* Any participant from whom Salmonella has been detected from at least two stool culture/PCR and 24hrs apart who has not received antibiotics by day 14 post-challenge
* Any participant in whom antibiotic use is felt to be clinically necessary (as decided by a medically qualified study doctor)

Follow up All participants will have to attend follow-up visits on day 28, 90, day 180, and day 365 where blood, saliva and stool samples will be taken. For safety reasons, pregnancy tests will be performed on female participants prior to the challenge and prior to starting antibiotics.

Vital signs, physical examination, blood and urine sampling, ECG, and mood assessment can be performed at any stage in the study if felt to be clinically indicated.

From these procedures, the study investigators will collect data including:

* the proportion of participants diagnosed with infection following challenge at different doses of the two challenge strains.
* safety and tolerability of challenge with the two strains of Salmonella Typhimurium (4/74 and D23580)
* the immune response following challenge which may correlate with protection from disease.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all the following criteria to be considered eligible for the study:

* Agree to give informed consent for participation in the study.
* Aged between 18 and 50 years inclusive at time of challenge.
* In good health as determined by medical history, physical examination, and clinical judgment of the study team.
* Agree (in the study team's opinion) to comply with all study requirements, including capacity to adhere to good personal hygiene and infection control precautions.
* Agree to allow his or her General Practitioner (and/or Consultant if appropriate), to be notified of participation in the study.
* Agree to allow study staff to contact his or her GP to access the participant's medical history and vaccination records.
* Agree to allow UKHSA and the local health protection unit to be informed of their participation in the study.
* Agree to give his or her close contacts written information informing them of the participant's involvement in the study and offer them voluntary screening for Salmonella carriage.
* Agree to a period of inpatient quarantine whilst symptomatic (In exceptional circumstances, the duration of inpatient quarantine may be extended.)
* Agree to have 24-hour contact with study staff during the four weeks post challenge and can ensure that they are contactable by mobile phone for the duration of the study period until antibiotic completion.
* Agree to allow the study team to hold the name and 24-hour contact number of a close friend, relative or housemate who will be kept informed of the study participant's whereabouts for the duration of the challenge period after quarantine (from the time of challenge until completion of antibiotic course). This person will be contacted if study staff are unable to contact the participant after discharge from inpatient quarantine.
* Have internet access to allow completion of the e-diary and real-time safety monitoring.
* Agree to avoid antipyretic/anti-inflammatory treatment from the time of challenge (Day 0) until advised by a study doctor or until 14 days after challenge.
* Agree to refrain from donating blood for the duration of the study.
* Agree to provide their National Insurance/Passport number for the purposes of Trial over-volunteering prevention system (TOPS) registration and for payment of reimbursement expenses.
* Participants must have received at least two doses of a SARS-CoV-2 vaccines that has been approved for use by the MHRA (or other national regulatory authority) four weeks prior to enrolment.
* Proficient in English at a level sufficient to understand, retain, weigh up and communicate the study details as outlined in the participant information sheet, in the opinion of the study investigator.

Exclusion Criteria:

The participant will not be enrolled if any of the following apply:

* History of microbiologically confirmed Salmonella infection.
* History of significant organ-specific and/or systemic disease that could interfere with trial conduct or completion. Including, for example, but not restricted to:

  * Cardiovascular disease, including specifically Atherosclerotic disease Stable or unstable angina Previous myocardial infarction Valvular heart disease Vascular disease, including specifically

    * Documented aneurysmal arterial disease
    * Peripheral arterial disease
    * Endovascular prosthesis oRespiratory disease
  * Haematological disease including sickle cell disease and sickle cell trait.
  * Endocrine disorders, including specifically diabetes mellitus
  * Renal or bladder disease, including history of renal calculi
  * Biliary tract disease, including specifically biliary colic, asymptomatic gallstones, or previous cholecystectomy
  * Gastro-intestinal disease including specifically, a current requirement for antacids, H2-receptor antagonists, proton pump inhibitors or laxatives OR Inflammatory bowel disease OR Confirmed diagnosis of irritable bowel syndrome as defined by the Rome IV criteria.
  * Neurological disease
  * Metabolic disease
  * Autoimmune disease
  * Psychiatric illness requiring hospitalisation
  * Known or suspected drug and/or alcohol misuse disorder
  * Chronic/Active Infectious disease including active tuberculosis
  * Severe infection requiring hospitalisation for intravenous antibiotics within the last 10 years. Exceptions to this would include a short course of intravenous antibiotics for appendicitis, biliary sepsis, diverticulitis, and cellulitis.
  * History of malaria infection within the past 12 months
  * History of joint replacement
  * History of any orthopaedic/osseous implanted prosthesis
  * Presence of other internal implanted device e.g. permanent pacemaker
* Have any known or suspected impairment of immune function, alteration of immune function, or prior immune exposure that may alter immune function to Salmonella infection resulting from, for example:

  * Congenital or acquired immunodeficiency, including IgA deficiency
  * Human Immunodeficiency Virus infection or symptoms/signs suggestive of an HIV-associated condition
  * Evidence of severe primary immunodeficiency, for example, severe combined immunodeficiency, Wiskott-Aldrich syndrome, and other combined immunodeficiency syndromes.
  * Currently being treated for malignant disease with immunosuppressive chemotherapy or radiotherapy, or who have received such treatment within at least the last six months
  * Individuals who have received a solid organ transplant and are currently on immunosuppressive treatment
  * Individuals who have received a bone marrow transplant, until within 12 months of finishing all immunosuppressive treatment,
  * Individuals receiving systemic high-dose steroids until at least three months after treatment has stopped.
  * Individuals receiving other types of immunosuppressive drugs (alone or in combination with lower doses of steroids) until at least six months after terminating such treatment.
  * Receipt of immunoglobulin or any blood product transfusion within 3 months of study start.
  * History of cancer (except squamous cell or basal cell carcinoma of the skin and cervical carcinoma in situ).
* Moderate or severe depression or anxiety as classified by the Hospital Anxiety and Depression Score at screening or challenge that is deemed clinically significant by the study doctors .
* Weight less than 50kg .
* Anyone taking long-term medication (e.g. analgesia, anti-inflammatories or antibiotics) that may affect symptom reporting or interpretation of the study results.
* Contraindication to cephalosporin, fluroquinolone, or macrolide antibiotics.
* Female participants who are pregnant, lactating or who are unwilling to ensure that they or their partner use effective contraception 30 days prior to challenge and continue to do so until two negative stool samples, a minimum of 3 weeks after completion of antibiotic treatment, have been obtained.
* Full-time, part-time, or voluntary occupations involving:

  * Clinical healthcare work
  * Social work with direct contact with young children (defined as those attending pre-school groups or nursery or aged under 2 years), or other clinically vulnerable children, adolescents
  * Clinical or social work with direct contact with highly susceptible patients or persons in whom Salmonella infection would have particularly serious consequences (unless willing to avoid work until demonstrated not to be infected with Salmonella in accordance with guidance from Public Health England and willing to allow study staff to inform their employer).
* Full time, part time or voluntary occupations involving:

  o Commercial food handling (involving preparing or serving unwrapped foods not subjected to further heating)
* Close household contact with:

  * Young children (defined as those attending pre-school groups, nursery or those aged less than 2 years)
  * Any individual who is immunocompromised.
  * Pregnant women
  * Household contacts aged over 70 years
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study period.
* Participants who have participated in another research study involving an investigational product that might affect risk of Salmonella infection or compromise the integrity of the study within the 30 days prior to enrolment (e.g. significant volumes of blood already taken in previous study) .
* Detection of any abnormal results from screening investigations, unless deemed not clinically significant.
* Any other social, psychological or health issues which, in the opinion of the study staff, may

  * Put the participant or their contacts at risk because of participation in the study,
  * Adversely affect the interpretation of the primary endpoint data,
  * Impair the participant's ability to participate in the study.
* Having previously received any experimental Salmonella vaccine as part of a clinical trial
* Have participated in previous Salmonella Typhi or Paratyphi challenge studies (with ingestion of challenge agent).
* Have a prolonged corrected QT interval (>450 milliseconds) on ECG screening
* Any employee of the sponsor or research site personnel directly affiliated with this study or their immediate family members.
* Inability to comply with any of the study requirements (at the discretion of the study staff).
* HLA-B27 positive

Temporary exclusion criteria at challenge

Participants will be temporarily excluded from challenge if presenting at the challenge visit with the following:

* Positive lateral flow test for SARS-CoV-2
* Significant acute or acute-on-chronic infection within the previous 7 days or have experienced fever (>37.5C) or subjective febrile symptoms within the previous 3 days.
* History of any antibiotic therapy during the previous 5 days.
* Any systemic corticosteroid (or equivalent) treatment in the previous 14 days, or for more than seven consecutive days within the past 3 months.
* Therapy with antacids, proton pump inhibitors or H2-receptor antagonists within 24 hours prior to challenge.
* Detection of gastrointestinal pathogens (other than Salmonella) in stool culture/PCR collected at the pre-challenge assessment (Day-7) including Shigella spp., Campylobacter spp., E. Coli O157, Giardia spp and Cryptosporidum spp, until two subsequent samples are negative. Detection of Salmonella spp. in stool prior to challenge (Day - 7) will result in exclusion from the study.
* Detection of Extended spectrum beta lactamase producing organisms or Carabapenem resistant organisms until two subsequent samples are negative.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The dose in CFU of Salmonella enterica subspecies enterica serovar Typhimurium (S. Typhimurium) 4/74 and D23580 strains required for 60-75% of volunteers to develop systemic Salmonellosis following oral challenge | Up to Day 14 post challenge (Inclusive)
  The proportion of participants who develop either:
  Fever ≥38°C on ≥2 occasions ≥12 hours apart AND/OR Salmonella Typhimurium bacteraemia

SECONDARY OUTCOMES:
The Salmonella colonisation rate following oral challenge with Salmonella Typhimurium 4/74 and D23580 strains at different doses | Up to Day 14 post challenge (Inclusive)
  The proportion from whom Salmonella Typhimurium is isolated from stool on ≥2 occasions ≥48 hours from challenge at different doses of each strain.
The Salmonella gastroenteritis rate following oral challenge of Salmonella Typhimurium 4/74 and D23580 strains at different doses. | Up to Day 14 post challenge (Inclusive)
  The proportion of participants at different doses at each strain developing Severe diarrhoea and/or Moderate diarrhoea plus Fever ≥38°C on ≥1 occasion and/or
  ≥1 Grade 2 gastrointestinal symptoms (abdominal pain, nausea, vomiting, tenesmus)
The persistent fever rate following oral challenge with Salmonella Typhimurium 4/74 and D23580 at different doses. | Up to Day 14 post challenge (Inclusive)
  The proportion of participants who develop fever ≥38°C on ≥2 occasions ≥12 hours apart at different doses of each strain.
The rate of systemic Salmonellosis according to an alternative composite diagnostic criterion following oral challenge of Salmonella Typhimurium 4/74 and D23580 at different doses. | Up to Day 14 post challenge (Inclusive)
  The proportion of participants meeting the criteria for a composite diagnosis of Salmonellosis at different doses of each strain defined as any of 1) Salmonella Typhimurium is isolated from stool on ≥2 occasions ≥48 hours from challenge and/or 2) Salmonella gastroenteritis and/or 3) fever ≥38°C on ≥2 occasions ≥12 hours apart and/or 4) Salmonella Typhimurium bacteraemia detected by blood culture and/or novel molecular methods
The safety of oral challenge with S. Typhimurium 4/74 and D23580 strains | Up to Day 14 post challenge (Inclusive)
  The proportion of participants at different doses of each strain reporting
  * Adverse events,
  * Adverse events of special interest,
  * SAEs,
  * SUSARs.
  * Concomitant medication usage as outlined in the study protocol
Clinical features following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  Solicited symptom profiles recorded in a diary card
Clinical features following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  Diarrhoea volume
Clinical features following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  Diarrhoea severity measures using a four point scale (Absent, Mild, Moderate, Severe)
Clinical features following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  The proportion of participants with any fever =>38C
Clinical features following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  The time to onset of first fever =>38C
Clinical features following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  Fever clearance time
Microbiological features of gastrointestinal infection following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  Time to onset in days in each group from challenge to first stool sample positive for Salmonella Typhimurium by culture and/or PCR
Microbiological features of gastrointestinal infection following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  magnitude of stool shedding measured in CFU/ml in quantitative stool culture analysis
Microbiological features of gastrointestinal infection following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  Duration of stool shedding in each group measured in days from first stool sample positive for Salmonella by culture and/or PCR
Microbiological features of bloodstream infection following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  The proportion of participants in each group developing any bacteraemia
Microbiological features of bloodstream infection following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  The duration of bacteraemia measured by time in hours from the first positive blood culture to first persistently negative blood culture
Microbiological features of bloodstream infection following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  Blood culture clearance time measured by time in hours from initiation of antibiotics treatment to first persistently negative blood culture
Microbiological features of bloodstream infection following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  Magnitude of bacteraemia measured in CFU/ml in quantitative blood culture samples collected immediately prior to the initiation of treatment
Microbiological features of bloodstream infection following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 14 post challenge (Inclusive)
  The time to onset of bacteraemia in each group, measured by hours since challenge
Biochemical and haematological laboratory parameters following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  Absolute values of laboratory parameters from time of challenge to Day 28 and/or Day 90, with specific reference to Total haemoglobin (d/L) Haemoglobin change from baseline (Hb g/l D0 - nadir Hb g/l) Total white cell count (x10e9/l) Neutrophil count (x10e9/l) Lymphocyte count (x10e9/l) Eosinophil count (x10e9/l) Monocyte/lymphocyte ratio Urea and electrolytes (Na+,K+, Urea, Creatinine - mmol/l) C-reactive protein (mg/l) Liver function tests (Bilirubin [umol/l], aspartate transaminase (AST IU/l), alkaline phosphatase (ALP IU/l), alanine transaminase (ALT IU/l), Albumin (g/l)
Serum antibody response following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  S. Typhimurium O-specific polysaccharide serum IgG and IgA concentration measured by ELISA
Serum antibody response following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  S. Typhimurium specific serum IgG and IgA concentration against other S. Typhimurium antigens measured by ELISA
Serum antibody response following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  Serum bactericidal antibody titres against Salmonella Typhimurium
Serum antibody response following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  S. Typhimurium specific antibody secreting cell and memory B-cell responses measured by ELISPOT
Serum antibody response following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  Other functional antibody activity measurements including systems serology platforms.
Mucosal antibody response following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains. | Up to Day 365 post challenge (Inclusive)
  S. Typhimurium specific IgG and IgA concentration measured by ELISA and other functional antibody activity measurements including systems serology platforms
Cell-mediated immune response following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  Lymphocyte sub-populations at baseline and following challenge as measured by flow cytometry and/or CyTOF
Cell-mediated immune response following oral challenge with S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  Frequency and magnitude of S. Typhimurium specific cell-mediated immune responses as measured by ELISPOT and flow cytometry and/or CyTOF

OTHER OUTCOMES:
To investigate how the human microbiota interacts with oral challenge of S. Typhimurium 4/74 or S. Typhimurium D23580 strains | Up to Day 365 post challenge (Inclusive)
  3.1 Pathogen specific and metagenomic analysis of stool and/or saliva to measure constituent microbiological flora (and their metabolome, transcriptome and anti-microbial resistance profile) at baseline and post-challenge time points
To investigate novel diagnostic methods for detecting S. Typhimurium infection | Up to Day 365 post challenge (Inclusive)
  Exploratory analysis of blood and faecal samples, including novel molecular techniques
To describe and compare additional host immune responses following oral challenge of S. Typhimurium 4/74 or S. Typhimurium D23580 strains. | Up to Day 365 post challenge (Inclusive)
  Analysis of B-cell repetoire, plasma cytokine profile and kinetics, additional exploratory immunology
To evaluate environmental contamination with Salmonella enterica in the near patient environment | Up to Day 365 post challenge (Inclusive)
  The pattern and proportion of environmental samples testing positive for Salmonella Typhimurium by culture or molecular methods
To evaluate host-pathogen interactions following Salmonella infection including the presence and mechanisms of Salmonella persister infected macrophages | Up to Day 365 post challenge (Inclusive)
  Exploratory analysis of infected immune cells from blood including, but not limited to, single-cell RNA-seq.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, England, United Kingdom

REFERENCES:
- [Derived] Smith C, Smith E, Rydlova A, Varro R, Hinton JCD, Gordon MA, Choy RKM, Liu X, Pollard AJ, Chiu C, Cooke GS, Gibani MM. Protocol for the challenge non-typhoidal Salmonella (CHANTS) study: a first-in-human, in-patient, double-blind, randomised, safety and dose-escalation controlled human infection model in the UK. BMJ Open. 2024 Jan 10;14(1):e076477. doi: 10.1136/bmjopen-2023-076477. PMID 38199617
- See also: Study website — https://www.imperial.ac.uk/infectious-disease/research/human-challenge/chants